CLINICAL TRIAL: NCT03127163
Title: Intrastromal Corneal Ring Was Effective for the Treatment of Mild Keratoconus
Brief Title: Intraestromal Corneal Ring in Mild Keratoconus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Mário Henrique Camargos de Lima, PhD, University of Sao Paulo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0591/11
Record Dates: First submitted 2017-04-12; First posted 2017-04-25 (Actual); Last update posted 2017-04-25 (Actual); Status verified 2017-04

CONDITIONS: Cornea; Eye Diseases; Keratoconus; Ophthalmological Disorder
MeSH Terms: conditions — Corneal Diseases; Eye Diseases; Keratoconus

STUDY DESIGN:
Intervention Model Description: Intraestromal corneal ring
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Mild Keratoconus (Other): A group of 65 patients with keratoconus who were implanted with an intrastromal corneal ring; the group was composed of 40 males (61.50%) and 25 females (38.50%), with a mean age of 27.88 ± 7.38 years (range, 17-47 years). The patients were fully informed about the study and signed a consent form previously approved by the ethics committee of our institution.
  We used the Amsler-Krumeich classification and included only patients classified as grade I or II. The investigators performed the intraestromal corneal ring surgery in the selected group.
  Interventions: Device: Intraestromal corneal ring

INTERVENTIONS:
Device: Intraestromal corneal ring — The patients underwent surgery to implant the intrastromal corneal ring (Ferrara Ophthalmics, Belo Horizonte, Brazil) using a manual technique. The procedures were performed by a single surgeon with extensive training in corneal surgery. All patients received the same ring, and the number (1 or 2 segments), thickness, and arc size were calculated using the nomogram provided by the manufacturer.
  Other Names: Ferrara ring

SUMMARY:
To determine whether the implantation of an intrastromal corneal ring is an effective treatment for a homogeneous group of mild keratoconus patients.

DETAILED DESCRIPTION:
A group of 65 patients with mild keratoconus were implanted with a Ferrara ring in a single eye. Six months after surgery, the aberrations were measured and the visual function was determined using clinical indices. The aberrations, especially comatic aberration (coma), were measured independently.

ELIGIBILITY:
Inclusion Criteria:

* Investigators used the Amsler-Krumeich classification and included only patients classified as grade I or II.

Exclusion Criteria:

* Investigators excluded patients with central corneal scarring, with other eye disorders, or with previous ocular surgery. We also excluded patients with a history of herpes infection, keratitis, corneal dystrophies, diagnoses of autoimmune diseases, systemic connective tissue disorders, or acute keratoconus.

Ages: 17 Years to 47 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 65 (Actual)
Dates: Start 2015-01-10 (Actual); Primary Completion 2016-01-10 (Actual); Study Completion 2017-01-10 (Actual)

PRIMARY OUTCOMES:
Aberrations were measured and the visual function was determined using clinical indices. | 3 months after surgery
  Wave front data

SECONDARY OUTCOMES:
UCVA | 3 months after surgery
  Uncorrected visual acuity
BCVA | 3 months after surgery
  Best corrected visual acuity

CONTACTS AND LOCATIONS:
Overall Officials: Mário Lima, PhD, Principal Investigator — São Paulo University investigator
Locations (1):
- Hospital das Clínicas, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No